CLINICAL TRIAL: NCT07079618
Title: A Randomized, Double-Blind, Placebo-Controlled, Single Ascending Dose Phase Ia Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetic Profile, Pharmacodynamics Profile, and Immunogenicity of SGC001 in Healthy Adult Subjects
Brief Title: A Research Study to Evaluate the Safety and Tolerability of SGC001 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Beijing Sungen Biomedical Technology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SG-SGC001-101
Record Dates: First submitted 2025-06-24; First posted 2025-07-23 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Anterior Myocardial Infarction
MeSH Terms: conditions — Anterior Wall Myocardial Infarction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SGC001 (Experimental): Administration should be initiated as early as possible, with a single intravenous injection completed within 6 hours of disease onset.
  Interventions: Drug: SGC001
- Placebo (Placebo Comparator): Administration should be initiated as early as possible, with a single intravenous injection completed within 6 hours of disease onset.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SGC001 — In this study, 6 dose groups are planned. 8 subjects are enrolled in each group. A total of 48 subjects will be enrolled. The administration method for each group is as follows: The drug SGC001 should be administered once via intravenous injection within 6 hours and the administration time 10 minutes.
  Arms: SGC001
Drug: Placebo — In this study, 6 dose groups are planned. 8 subjects are enrolled in each group. A total of 48 subjects will be enrolled. The administration method for each group is as follows: The drug placebo should be administered once via intravenous injection within 6 hours and the administration time 10 minutes.
  Arms: Placebo

SUMMARY:
Acute Myocardial Infarction (AMI) is an acute ischemic necrosis that occurs following acute stenosis or occlusion of the coronary arteries, and it is associated with a high morbidity and mortality rate. Acute myocardial infarction typically occurs in middle-aged and elderly individuals, according to the American Heart Association, with the average age of first occurrence being 65.1 years for men and 72.0 years for women. Myocardial infarction (MI) has a significant impact on global health, affecting over 7 million people worldwide annually. In addition, MI can impose a substantial economic burden on society and families. The research study is a Randomized, Double-Blind, Placebo-Controlled, Single Ascending Dose Phase Ia Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetic Profile, Pharmacodynamics Profile, and Immunogenicity of SGC001 in Healthy Adult Subjects

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who fully understand the purpose, nature, method, and potential adverse reactions of the trial, and who voluntarily sign the informed consent form and agree to participate in the study.
2. Healthy male or female subjects aged 18 ~ 50 years (both inclusive, based on the time of signing the informed consent form).
3. Body mass index (BMI): 19.0 ~ 26.0 kg/m2 (both inclusive), body weight of male subjects ≥50.0 kg, and body weight of female subjects ≥45.0 kg.
4. Female subjects of childbearing potential must agree to use effective contraception from screening until 3 months after receiving the investigational drug. In addition, they must agree to refrain from collecting or donating eggs during this period; their male partner of childbearing potential must also agree to use effective contraception during this period.
5. Male subjects of childbearing potential must agree to use effective contraception and have no plans to conceive or donate sperm from screening until 3 months after receiving the investigational drug. During this period, their female partner of childbearing potential must also agree to use effective contraception.

Exclusion Criteria:

1. Individuals with known allergy to therapeutic protein drugs or food or who may be allergic to the test drug or any component of the investigational drug, based on the investigator's judgment.
2. Individuals with a history of cardiovascular disease.
3. Individuals with a history of acute or chronic bronchospasm, including treated or untreated asthma, and chronic obstructive pulmonary disease (COPD).
4. Individuals with a history of autoimmune disease.
5. Individuals with a history of malignant tumors.
6. Individuals with clinically significant abnormalities on physical examination, vital signs examination, electrocardiogram or laboratory tests, as judged by the clinician.
7. Individuals with a history of drug abuse within the past 5 years, the presence of drug abuse within 3 months before the study, or a positive drug abuse screening result.
8. Individuals who have smoked within 3 months before screening (consuming ≥ 5 cigarettes per day) or habitual use of nicotine containing products.
9. Individuals who have consumed more than 14 units of alcohol per week (1 unit of alcohol = 360 mL of beer or 45 mL of spirits with 40% of alcohol content or 150 mL of wine) within 3 months prior to screening, or who consume alcohol-containing products within 48 hours before dosing, or who have a positive alcohol breath test result at screening and/or D-1.
10. Individuals who have received monoclonal antibody or biologic therapy within 3 months prior to receiving the investigational drug.
11. Individuals who have received medications that may affect the immune system (e.g., immunosuppressants, cytokines and cytokine inducers,) within 3 months prior to receiving the investigational drug.
12. Individuals who have received anticoagulant or antiplatelet medications within 28 days prior to receiving the investigational drug.
13. Individuals who have received any vaccine within 28 days prior to receiving the investigational drug, or who plan to receive a vaccine during the trial period.
14. Individuals who have suffered from clinically significant major diseases or undergone major surgical procedures within 28 days prior to receiving the investigational drug, or who anticipate requiring major surgery during the trial period.
15. Individuals who have used any prescription drugs, over-the-counter drugs, Chinese herbal medicines, or health supplements within 14 days prior to receiving the investigational drug or within the 5 half-lives of the drug (whichever is longer).
16. Individuals whose screening viral serology tests are positive for human immunodeficiency virus antigen/antibodies (HIV-Ag/Ab), hepatitis B surface antigen (HBsAg), hepatitis C virus antibodies (HCV-Ab), or antibodies to Treponema pallidum (TP-Ab).
17. Individuals who have difficulty in venous blood collection or have a history of needle and blood fainting.
18. Women who have positive result in pregnancy test or are breastfeeding at Screening or D-1.
19. Individuals who have participated in other drug clinical studies and received other clinical trial drugs within 3 months prior to receiving the investigational drug.
20. Individuals who have history of blood donation or massive blood loss (≥ 400 mL) within 3 months prior to screening.
21. Any other circumstance that, in the judgement of the investigator, may affect the ability of the subject to provide informed consent or to follow the trial protocol, or where the subject's participation in the trial may affect the outcome of the trial or his/her safety.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2024-08-20 (Actual); Primary Completion 2025-07-15 (Actual); Study Completion 2025-07-15 (Actual)

PRIMARY OUTCOMES:
Adverse events (AEs) | From randomisation to end-of-study (up to 57 days)
  Adverse events (AEs)
Serious adverse events (SAEs) | From randomisation to end-of-study (up to 57 days)
  Serious adverse events (SAEs)
ECG QT Interval | From randomisation to end-of-study (up to 57 days)
  ECG QT Interval
Number of participants with Laboratory tests | From randomisation to end-of-study (up to 57 days)
  hematology, blood chemistry, urinalysis, and coagulation

SECONDARY OUTCOMES:
Maximum Concentration (Cmax) | Day 1-Day 4, Day 6, Day 8-Day 57
  Maximum Concentration (Cmax)
Time to maximum concentration (Tmax) | Day 1-Day 4, Day 6, Day 8-Day 57
  time to maximum concentration (Tmax)
Area under the plasma concentration-time curve from time 0 to the last quantifiable time point postdose (AUC0-t) | Day 1-Day 4, Day 6, Day 8-Day 57
  Area under the plasma concentration-time curve from time 0 to the last quantifiable time point postdose (AUC0-t)
Area under the plasma concentration-time curve from time zero to infinity (AUC0-inf) | Day 1-Day 4, Day 6, Day 8-Day 57
  Area under the plasma concentration-time curve from time zero to infinity (AUC0-inf)
Elimination half-life (t1/2) | Day 1-Day 4, Day 6, Day 8-Day 57
  Elimination half-life (t1/2)
Elimination rate constant (λz) | Day 1-Day 4, Day 6, Day 8-Day 57
  Elimination rate constant (λz)
Interleukin-6(IL-6) [PD endpoints] | Day 1-Day 2,Day 4,Day 8-Day 22
  Interleukin-6(IL-6)
Tumor necrosis factor-α（TNF-α)[PD endpoints] | Day 1-Day 2,Day 4,Day 8-Day 22
  Tumor necrosis factor-α（TNF-α)
Immunoglobulin G (IgG)[PD endpoints] | Day 1-Day 2,Day 4,Day 8-Day 22
  Immunoglobulin G (IgG)
Interleukin-1 β (IL-1 β)[PD endpoints] | Day 1-Day 2,Day 4,Day 8-Day 22
  Interleukin-1 β (IL-1 β)
Qualitative detection of anti-drug antibodies in serum（Anti-drug antibody (ADA)） | Day 1,Day 8-Day 15,Day 29-Day 57
  Qualitative detection of anti-drug antibodies in serum, followed by calculation of the positivity rate as the number of positive samples divided by the total number of samples

CONTACTS AND LOCATIONS:
Overall Officials: Yang Lin, Ph.D, Principal Investigator — Beijing Anzhen Hospital
Locations (1):
- Beijing Anzhen Hospital Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
The individual participant data(IPD) will be shared if necessary